CLINICAL TRIAL: NCT03106649
Title: Echocardiography Based Algorithm for Prevention and Treatment of Spinal Hypotension- A Prospective Randomised Controlled Study
Brief Title: Echocardiography Based Algorithm for Spinal Anaesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Dr. SUNDARA KANNAN, PRINCIPAL INVESTIGATOR, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10306/PG-2Trg/2015/1696
Record Dates: First submitted 2017-03-29; First posted 2017-04-10 (Actual); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Hypotension
MeSH Terms: conditions — Hypotension | interventions — Echocardiography

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gr (E) (Experimental): The group in which the proposed algorithm for prevention and treatment of spinal hypotension will be tested with regard to fluid and vasopressor use, by means of echocardiography.
  Interventions: Device: Echocardiography; Device: Treatment of spinal hypotension
- Gr (S) (No Intervention): The control group in which the anesthesia (fluid and vasopressor) management will be decided by the attending anesthesiologist

INTERVENTIONS:
Device: Echocardiography — Before administration of spinal anesthesia, Echocardiography will be performed to determine the LVEDA. If the LVEDA is more than 10 square cms, the patient will be considered as volume replete and spinal anesthesia will be administered. If the LVEDA is less than 10 square cms, a fluid bolus of 250 ml of a balanced salt solution will be given and LVEDA reassessed. This will be repeated till the LVEDA is more than 10 square cms or fluid bolus has been given twice and still the LVEDA is less than 10 square centimeters, in which case phenylephrine 1-2µg/kg will be given before administering spinal anesthesia.
  Arms: Gr (E)
Device: Treatment of spinal hypotension — For treatment of spinal hypotension, in the event of hypotension(defined as a mean arterial pressure less than 60 mm Hg or decrease in mean arterial pressure of more than 20% from the baseline value) after spinal anesthesia, the LVEDA will be assessed. If more than 10 square centimeters, the patient will be considered volume replete and a vasopressor in the form of phenylephrine 1-2µg/kg will be given. If the LVEDA is less than 10 square centimeters, a volume bolus of 250ml will be given. On reassessment if the LVEDA is still less than 10 square centimeters the volume bolus can be repeated. In the event of hypotension persisting in spite of volume resuscitation, phenylephrine 1-2µg/kg will be given.
  Arms: Gr (E)

SUMMARY:
The main aim of the study is to compare the proposed algorithm for preventing and treating spinal hypotension with normal anesthesia management of a spinal anesthesia.

The proposed algorithm mainly will depend upon the left ventricular end diastolic area measurement by transthoracic echocardiography to assess the left ventricular preload status and its usefulness in preventing and treating spinal hypotension.

DETAILED DESCRIPTION:
Aims and Objectives:

Primary aim:

To compare an echocardiography based algorithm of hemodynamic management as compared to standard practice in decreasing the incidence of spinal hypotension (number of patients developing a decrease in MAP >20% of baseline or MAP <60 mm Hg).

Secondary aims:

1. To compare the number of episodes, magnitude of hypotension (lowest value of BP) and duration of hypotension in either group.
2. To compare the amount of fluids and vasopressors administered to maintain hemodynamic stability in either group.

MATERIALS AND METHODS:

This study is designed as prospective, randomized intention to treat trial. After obtaining written informed consent, a total of 60 patients, above 40 years of age presenting for elective lower abdominal or lower limb surgery and eligible to receive a subarachnoid block at the Postgraduate Institute of Medical Education and Research, Chandigarh from 1st January 2016 to March 31st 2017 will be enrolled in this study. Patients with contraindications to a central neuraxial block such as pre- existing coagulopathy, local sepsis at site of insertion, ongoing hemodynamic instability (defined as systolic blood pressure< 90 mm Hg or MAP< 65mm Hg), unwillingness to undergo a regional anesthesia, co- existing pregnancy, spinal dysraphism or, previous history of spinal instrumentation or surgery, chest deformity, demonstrated systolic dysfunction on screening echocardiography (defined as left ventricular ejection fraction <50% or, fractional shortening < 25%), valvular heart disease (known or diagnosed on screening echocardiography), chronic renal or liver disease and unwilling to participate in the trial will be excluded.

After standard preoperative fasting of 8hr, all patients will receive intravenous access and non-invasive blood pressure monitor set to be recorded automatically every 2 minutes, five lead continuous electrocardiography, pulse oximetry, and capnography for non-intubated patients inside OR. In addition, a screening echocardiogram for right and/ or left heart dysfunction (fractional shortening< 25% or ejection fraction < 50%/ and tricuspid annular plane systolic excursion < 17 mm) and exclusion of valvular heart disease will be performed. If an abnormality is detected patient will be excluded from the study at this point, enrolment proceeding on an intention to treat basis.

Thereafter the patients will be randomized into either of two groups using computer generated random number and sealed envelope method: Gr (E) echocardiography based fluid and hemodynamic management or, Gr (S) standard anaesthetic management. In group E patients, before administering spinal anesthesia, a transthoracic echocardiography (TTE) will be performed to determine the LVEDA using the mid papillary parasagittal short axis (PSAX) view. The average of at least 3 LVEDA measured on above view by an experienced anesthesiologist in TTE will be used for fluid management, as per the proposed algorithm . If spinal hypotension does occur in patients in group E, it will be managed according to the same proposed algorithm.

THE PROPOSED ECHOCARDIOGRAPHY BASED ALGORITHM :

The left ventricular end diastolic area (LVEDA) will be measured by Transthoracic echocardiography using the parasternal short axis view. If the LVEDA is more than 10 square centimeters, the left ventricular preload status will be deemed adequate and administration of spinal anesthesia will be proceeded as usual. If the LVEDA is less than 10 square cms, a fluid(NS/Balanced salt solution) bolus of 250 ml will be administered and LVEDA reassessed. If more than 10 square cms, spinal anaesthesia will be administered. If less, a second bolus of 250 ml fluid will be given and then LVEDA reassessed. If more than 10 square centimeters, spinal anaesthesia will be administered, if not the patient will be considered fluid unresponsive and spinal anesthesia will be administered after giving a phenylephrine iv bolus of 1-2µg/kg and then spinal anaesthesia administered. In the event of postspinal hypotension within 30 minutes of giving spinal anaesthesia, the LVEDA will be reassessed. If more than 10 square centimeters, volume status will be considered adequate and patient will be given a vasopressor bolus of 1-2µg/kg of phenylephrine. If less than 10 square centimeters, the patient volume status will be considered low and a fluid bolus of 250ml and LVEDA reassessed and managed as in a prespinal LVEDA of less than 10 square centimeters.

The patients in group S will receive fluid and vasopressor therapy (if required) as deemed appropriate by the attending anaesthesiologist. The attending anaesthesiologist will be will target a MAP, such that it does not fall below 60 mm Hg nor below >20% of its baseline value.

The anaesthetic management protocol will be standardized for both the groups namely all patient will receive 3.0ml of local anaesthetic fentanyl mixture [2.5ml of 0.5%bupivacaine + 0.5ml(25µg) of fentanyl], ringer lactate/ any balanced salt solution(BSS) for fluid management and phenylephrine 1-2µg/kg intermittent boluses to treat hypotension. No i.v sedative or analgesic medication will be administered until completion of study. Patient position will be kept supine till end of the study period and surgical incision will be given thereafter. The attending anesthesiologist managing case will be not be involved in the study and will be blinded for the goal and parameters recorded in the study.

The patient demographic data characteristics such as age, sex, height, weight, observed echocardiographic parameters, LVEDA and changes in LVEDA following bolus volume administration will be noted. The echocardiographic parameters will be recorded for later analysis. The hemodynamic parameters will be recorded for every 1 minutes for 1st 10 minutes of spinal drug administration and thereafter at 5 minutes interval till the study period. The number of episodes of hypotension and the total fraction of time spent below target values in the first 30 minutes post spinal block (defined by decrease in MAP exceeded >20% from baseline and absolute value <60 mm Hg), magnitude of hypotension (lowest value of BP), volume of crystalloid / colloid, number of times vasopressors were used and total doses of vasopressors required will be noted. Any side effect like nausea/ vomiting, persistent hypotension defined by decrease in MAP exceeding >20% from baseline for 5 minutes or more will be noted.

The blood pressure values within 30 minutes of administering spinal anesthesia will be considered and analysed for study purposes, to exclude the effect of surgical factors on hemodynamics.

ELIGIBILITY:
Inclusion Criteria:

- above 40 years of age presenting for elective lower abdominal or lower limb surgery and eligible to receive a subarachnoid block.

Exclusion Criteria:

* . Patients with contraindications to a central neuraxial block such as pre- existing coagulopathy, local sepsis at site of insertion, ongoing hemodynamic instability (defined as systolic blood pressure< 90 mm Hg or MAP< 65mm Hg), unwillingness to undergo a regional anaesthesia, co- existing pregnancy, spinal dysraphism or, previous history of spinal instrumentation or surgery, chest deformity, demonstrated systolic dysfunction on screening echocardiography (defined as LVEF <50% or, fractional shortening < 25%), valvular heart disease (known or diagnosed on screening echo), chronic renal or liver disease and unwilling to participate in the trial.

Min Age: 40 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-04 (Actual); Primary Completion 2017-05 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of hypotension | 30 minutes
  To compare an ECHO based algorithm of hemodynamic management as compared to standard practice in decreasing the incidence of post spinal hypotension (MAP >20% of baseline or MAP <60 mm Hg).

SECONDARY OUTCOMES:
number of episodes of hypotension. | 30 minutes
  To compare the number of episodes of hypotension in either group.
magnitude of hypotension. | 30 minutes
  To compare the magnitude of hypotension (lowest value of BP) in either group.
duration of hypotension. | 30 minutes
  To compare the duration of hypotension (in minutes) in either group.
use of IV fluids | 30 minutes
  To compare the amount of fluids(milliliters) administered to maintain hemodynamic stability in either group.
use of vasopressors | 30 minutes
  To compare the amount of vasopressors (micrograms/kg) administered to maintain hemodynamic stability in either group.

CONTACTS AND LOCATIONS:
Overall Officials: Sundara Kannan, MBBS, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh; Bhupesh Kumar, MBBS,MD,DM, Study Chair — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- Postgraduate Institute of Medical Education and Research, Chandigarh, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No